CLINICAL TRIAL: NCT02770794
Title: Multicenter Prospective Trial to Investigate Accuracy of Ultrasound to Predict Relapse After Discontinuation of Infliximab and Efficacy/Safety of Readministration of Infliximab in Patients With Rheumatoid Arthritis in Low Disease Activity
Brief Title: Optimization of Infliximab Withdrawal Strategy for Rheumatoid Arthritis
Acronym: OPTIWIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chiba University (Other)
Responsible Party: Principal Investigator, Kei Ikeda, Senior Lecturer, Chiba University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 137
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Masking Description: Investigators were masked for ultrasound results
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): Discontinue infliximab; Receive infliximab when relapse
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Discontinue infliximab; receive Infliximab when relapse

SUMMARY:
This multicenter prospective clinical trial investigates the accuracy of ultrasound to predict relapse after discontinuation of infliximab and the efficacy/safety of readministration of infliximab in patients with rheumatoid arthritis in a low disease activity state.

DETAILED DESCRIPTION:
The objective of this multicenter prospective clinical trial is to determine whether ultrasound predicts relapse after discontinuation of infliximab more accurately than does clinical index and to investigate the efficacy and safety of restarting infliximab after relapse in patients with rheumatoid arthritis in remission or low disease activity on infliximab treatment. Infliximab is discontinued in all enrolled patients. Patients are followed up for 48 weeks for monitoring relapse. If relapse occurs, patients receive readministration of infliximab and are further followed up for 24 weeks to determine the efficacy and safety of infliximab readministration. Primary endpoint is the difference in area under curve (AUC) of receiver operator characteristics (ROC) analysis between total power Doppler score and Disease Activity Score (DAS) 28 at baseline to predict relapse within 48 weeks after discontinuation of infliximab.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. RA patients who fulfill 2010 ACR/EULAR Classification Criteria
3. Patients who have been treated with infliximab (Remicade) for 26 weeks or longer
4. DAS28 (CRP) < 3.2 at screening
5. Patients who give written informed consent after receiving sufficient information -

Exclusion Criteria:

1. Receiving prednisolone > 10 mg/day
2. Receiving biological or molecular-target anti-rheumatic drug
3. Alteration of the dose of corticosteroid or anti-rheumatic drug within 8 weeks prior to screening visit
4. Alteration of the dose of non-steroid anti-inflammatory drug within 4 weeks prior to screening visit
5. History of infusion reaction to infliximab
6. Current infection which requires treatment
7. Current or previous demyelinating disorder
8. Current congestive heart failure which requires treatment
9. Breast-feeding or pregnant/possibly pregnant woman, or woman who does not agree to prevent conception during and 6 months after study period
10. Patients whom investigator or co-investigator consider inappropriate for other reasons -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Area under the Receiver Operator Characteristic (ROC) curve for total power Doppler score to predict relapse | 48 week
  Area under the ROC curve for total power Doppler score at baseline to predict relapse within 48 weeks after discontinuation of infliximab

SECONDARY OUTCOMES:
Area under the ROC curve for total gray-scale score to predict relapse | 48 week
  Area under the ROC curve for total gray-scale score at baseline to predict relapse within 48 weeks after discontinuation of infliximab
Change in van der Heijde modified Sharp score | 48 week
  Change in van der Heijde modified Sharp score at 48 week
Change in Health Assessment Questionnaire-Disability Index | 48 week
  Change in Health Assessment Questionnaire-Disability Index at 48 week
Change in EuroQoL 5 dimensions-5L | 48 week
  Change in EuroQoL 5 dimensions-5L at 48 week
EULAR response criteria based on DAS28 after readministration of infliximab | 12 week after relapse
  EULAR response criteria based on DAS28 at 12 week after relapse and readministration of infliximab
Number of adverse events as assessed by CTCAE v4.0 | Through study completion, an average of 60 weeks
  Number of adverse events as assessed by CTCAE v4.0 through study completion, an average of 60 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chiba University Hospital, Chiba, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iwamoto T, Ikeda K, Hosokawa J, Yamagata M, Tanaka S, Norimoto A, Sanayama Y, Nakagomi D, Takahashi K, Hirose K, Sugiyama T, Sueishi M, Nakajima H. Prediction of relapse after discontinuation of biologic agents by ultrasonographic assessment in patients with rheumatoid arthritis in clinical remission: high predictive values of total gray-scale and power Doppler scores that represent residual synovial inflammation before discontinuation. Arthritis Care Res (Hoboken). 2014 Oct;66(10):1576-81. doi: 10.1002/acr.22303. PMID 24515410
- [Background] Tanaka Y, Takeuchi T, Mimori T, Saito K, Nawata M, Kameda H, Nojima T, Miyasaka N, Koike T; RRR study investigators. Discontinuation of infliximab after attaining low disease activity in patients with rheumatoid arthritis: RRR (remission induction by Remicade in RA) study. Ann Rheum Dis. 2010 Jul;69(7):1286-91. doi: 10.1136/ard.2009.121491. Epub 2010 Apr 1. PMID 20360136